CLINICAL TRIAL: NCT01160692
Title: A Randomized, Placebo-controlled, Parallel Group, Double Blind Study to Evaluate the Cognitive Effects and Tolerance of a Multi-Vitamin/Mineral Preparation Containing Gingko in Elderly Subjects With Age Associated Memory Impairment
Brief Title: A Study to Evaluate The Effects Of a Multivitamin/Mineral With Ginko In Subjects With Age Associated Memory Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11954
Record Dates: First submitted 2009-10-08; First posted 2010-07-12 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2010-07

CONDITIONS: Age-Related Memory Disorders
Keywords: Memory; Cognitive Function; Elderly; Gingko; Age Associated Memory Impairment (AAMI)
MeSH Terms: conditions — Memory Disorders | interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Dietary Supplement: Multivitamin/Multimineral/Ginkgo (BAY 81-2775)
- Arm 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Multivitamin/Multimineral/Ginkgo (BAY 81-2775) — Multivitamin/Multimineral/Ginkgo (BAY 81-2775), daily oral intake of film coated tablets for 3 months
  Arms: Arm 1
Other: Placebo — Daily oral intake of matching placebo tablets for 3 months
  Arms: Arm 2

SUMMARY:
A Study to evaluate the cognitive effects and tolerance of a Multi-Vitamin/Mineral Preperation containing Gingko in elderly subjects with age associated memory impairment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is generally healthy (includes subjects presenting with mild chronic diseases where the disease and/or the pharmacological treatment does not result in psychomotor impairment or improvement).
* Subject is of either gender, and 60+ years of age, inclusive.
* Subject demonstrates Age Associated Memory Impairment after completion of the CDR test battery and comparison to normative data.
* Female subject who is post-menopausal.
* Subject is able to understand the study instructions and has given written informed consent prior to study participation.
* Subject admitted to this study is oriented to person, place and time and has the ability to communicate with the study staff.
* Subject is, in the opinion of the study staff, motivated to participate and complete the study as instructed.
* Subject is willing to be attend visits in a well-rested state.

Exclusion Criteria:

* Subject has participated in an interventional study within the one month prior to screening.
* Intake within three months prior to screening, or intended intake during the study, of one of the following: Ginkgo biloba, St John's Wort, Ginseng, Gotu Kola (Indian Pennywort), or daily doses of vitamin E (-tocopherol) above 30 mg, folic acid above 400 g, vitamins B-1 (thiamine), B-2 (riboflavin), B-6 (pyridoxine) above 2 mg, or other cognition enhancers.
* Subject has a history of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
* Subject has a history of Alzheimers disease, dementia, mental retardation, Morbus Parkinson, or any other mental disorders.
* Subject has not been diagnosed with AAMI after completion of the CDR test battery and comparison to normative data.
* Subject has a history of any bleeding/coagulation disorder (e.g., haemophilia, Protein C or S deficiency).
* Subject is taking/being treated with a concomitant medication which may affect/inhibit blood coagulation (e.g., warfarin, aspirin, heparin).
* Subject has history of relevant vascular disorders (e.g., carotid stenosis, stroke, PRIND, coronary artery disease, peripheral vascular disease, thrombosis).
* Subject has Body Mass Index (BMI) above 40 kg/m2 (severely obese).
* Subject smokes more than 15 cigarettes, or equivalent daily.
* Subject has moderate-to-severe hepatic impairment.
* Subject has history of alcohol or drug abuse.
* Subject has known allergies or intolerance to any ingredients in the study preparations.
* Subject is intending to undergo surgery during or immediately upon completion (within two weeks) of study participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The effect of the multi-vitamin/-mineral preparation containing gingko on major aspects of human cognitive function employing a computerized cognitive assessment system. | From baseline up to 12 weeks

SECONDARY OUTCOMES:
The effects of the multi-vitamin/-mineral preparation containing gingko on subjective memory using questionnaires. | From baseline up to 12 weeks
Tolerance of the daily oral intake of the multi-vitamin/-mineral preparation containing gingko. | From baseline up to 14 weeks
The effects of the multi-vitamin/-mineral preparation containing gingko on mood using questionnaires. | From baseline up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Newcastle upon Tyne, United Kingdom